CLINICAL TRIAL: NCT03633396
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind, Multiple Dose Study to Evaluate the Efficacy and Safety of ANB019 in Subjects With Palmoplantar Pustulosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Imsidolimab (ANB019) in Adults With Palmoplantar Pustulosis
Acronym: POPLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANB019-003; 2017-004022-15 (EudraCT Number)
Record Dates: First submitted 2018-07-19; First posted 2018-08-16 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2022-05

CONDITIONS: Palmoplantar Pustulosis
Keywords: PPP
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo administered by subcutaneous injection on Day 1 followed by monthly doses of placebo by subcutaneous injection on Days 29, 57, and 85.
  Interventions: Drug: Placebo
- imsidolimab (Experimental): Participants will receive 200 mg imsidolimab by subcutaneous injection on Day 1 followed by monthly doses of 100 mg imsidolimab by subcutaneous injection on Days 29, 57, and 85.
  Interventions: Biological: Imsidolimab

INTERVENTIONS:
Biological: Imsidolimab — Administered by subcutaneous injection once a month
  Other Names: ANB019
  Arms: imsidolimab
Drug: Placebo — Administered by subcutaneous injection once a month
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy and safety, and pharmacokinetic (PK) profile of multiple doses of imsidolimab (ANB019) in adults with palmoplantar pustulosis (PPP)

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of PPP
* Disease duration of at least 6 months prior to screening
* Present with active pustules on palms or/and soles at screening

Exclusion Criteria:

* Any other ongoing inflammatory disease that interfere with the investigator's ability to evaluate the subject's response to therapy
* History of recurrent or active/serious infection
* Ongoing use of psoriasis prohibited medication

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (18):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Encino, California
  - Investigational Site, Santa Monica, California
  - Investigational Site, Fort Lauderdale, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Pembroke Pines, Florida
  - Investigational Site, Tampa, Florida
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Plainfield, Indiana
  - Investigational Site, Overland Park, Kansas
  - Investigational Site, Ann Arbor, Michigan
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Wilmington, North Carolina
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Norman, Oklahoma
  - Investigational Site, Portland, Oregon
  - Investigational Site, Dallas, Texas
- Canada (5):
  - Investigational Site, Surrey, British Columbia
  - Investigational Site, Greater Sudbury, Ontario
  - Investigational Site, Markham, Ontario
  - Investigational Site, Drummondville, Quebec
  - Investigational Site, Montreal, Quebec
- Germany (5):
  - Investigational Site, Bad Bentheim
  - Investigational Site, Berlin
  - Investigational Site, Bonn
  - Investigational Site, Hamburg
  - Investigational Site, Schwerin
- Poland (8):
  - Investigational Site, Gdansk
  - Investigational Site, Katowice
  - Investigational Site, Lodz
  - Investigational Site, Olsztyn
  - Investigational Site, Ostrowiec Świętokrzyski
  - Investigational Site, Rzeszów
  - Investigational Site, Szczecin
  - Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this trial at 36 sites located within North America and Europe.
Pre-assignment Details: Participants were randomized equally to one of two treatment groups. Randomization was stratified based on the participant's history of plaque psoriasis, to ensure that the number of participants enrolled with plaque psoriasis did not exceed 50%.
Groups:
- Placebo: Participants received placebo administered by subcutaneous injection on Day 1 followed by monthly doses on Days 29, 57, and 85.
- Imsidolimab: Participants received 200 mg imsidolimab by subcutaneous injection on Day 1 followed by monthly doses of 100 mg imsidolimab by subcutaneous injection on Days 29, 57, and 85.
Period: Overall Study
Arm/Group | Placebo | Imsidolimab
Started | 29 | 30
Completed | 23 | 24
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Coronavirus Disease 2019 (COVID-19) Restrictions | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set (all randomized participants)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Imsidolimab | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.59) | 52.3 (12.10) | 50.1 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 26 | 30 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 1 | 4
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Palmoplantar Pustulosis Psoriasis Area Severity Index Score [Mean (Standard Deviation); unit: score on a scale] — The Palmoplantar Pustulosis Area and Severity Index (PPPASI) is used to assess the severity of palmoplantar pustulosis lesions. The glabrous skin of both palms and both soles are assessed for erythema, pustules and desquamation (scaling), each on a scale from 0 (none) to 4 (very severe). The area affected of each palm and sole is scored from 0 (0%) to 6 (90-100%). The PPPASI total score ranges from 0 to 72. A higher score indicates more severe disease.
  score on a scale | 19.47 (11.633) | 16.18 (8.045) | 17.80 (10.022)
History of Plaque Psoriasis [Count of Participants; unit: Participants]
  Yes | 7 | 7 | 14
  No | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Palmoplantar Pustulosis Psoriasis Area Severity Index (PPPASI)
Description: The Palmoplantar Pustulosis Area and Severity Index (PPPASI) is used to assess the severity of palmoplantar pustulosis lesions and their response to therapy. The glabrous skin of both palms and both soles are assessed for erythema, pustules, and desquamation (scaling), each on a scale from 0 (none) to 4 (very severe). The area affected of each palm and sole is scored from 0 (0%) to 6 (90-100%). Scores for the 3 characteristics of PPP are summed and adjusted for the area affected, and the scores for each palm and sole are added to calculate the total score. The PPPASI total score ranges from 0 to 72. A higher score indicates more severe disease, and a negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 16
Population: Intent-to-treat analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Imsidolimab
Number analyzed (Participants) | 24 | 24
score on a scale | -6.0 (1.48) | -6.1 (1.46)
Statistical Analysis 1: Comparison: Placebo vs Imsidolimab; The change from Baseline in PPPASI at Week 16 was analyzed using a a general linear mixed model for repeated measures (MMRM). The model included fixed effects for treatment, history of plaque psoriasis (Yes/No), visit, treatment by visit interaction, and Baseline PPPASI score as covariate; Test type: Other; p = 0.944, Mixed-model Repeated Measures (MMRM); MMRM including fixed effects of treatment, history of plaque psoriasis, visit, treatment by visit interaction, and Baseline PPPASI score as covariate; Least Squares (LS) Mean Difference = -0.1, 95% CI 2-sided [-4.05 to 3.77], Standard Error of Mean 1.98 — Least-squares mean difference = Imsidolimab - Placebo

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Clinical safety was evaluated by reporting incidence of adverse events up to week 24. TEAEs are defined as new events that occured during or after first dose of study drug or any event that worsens after first dose of study drug.
  A serious AE (SAE) is defined as any untoward medical occurrence that resulted in death, was life-threatening, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or an important medical event that may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed above.
  Severity was assessed by the Investigator as mild (easily tolerated, causing minimal discomfort and not interfering with everyday activities), moderate (causes sufficient discomfort and interferes with normal everyday activities) or severe (prevents normal everyday activities).
  The Investigator assessed the relationship between study treatment and each AE based on clinical judgement.
Time Frame: From first dose of any study drug to Week 24
Population: Safety Analysis Set (all randomized participants who received at least 1 dose of imsidolimab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Imsidolimab
Number analyzed (Participants) | 29 | 30
Participants
  Any treatment-emergent adverse event (TEAE) | 20 | 21
  TEAE related to study drug | 3 | 6
  Severe TEAE | 1 | 0
  Serious TEAE | 1 | 0
  TEAE of special interest | 1 | 0
  TEAE leading to discontinuation of study treatment | 2 | 1
  TEAE leading to study discontinuation | 1 | 1
  TEAE leading to death | 0 | 0
  TEAE related to injection site reaction | 0 | 0
  Disease related TEAE | 6 | 2

3. Secondary Outcome: Percentage of Participants Who Achieved 50% Reduction (Improvement) From Baseline in Palmoplantar Pustulosis Psoriasis Area Severity Index Score (PPPASI 50)
Description: The Palmoplantar Pustulosis Area and Severity Index (PPPASI) is used to assess the severity of palmoplantar pustulosis lesions and their response to therapy. The glabrous skin of both palms and both soles are assessed for erythema, pustules, and desquamation (scaling), each on a scale from 0 (none) to 4 (very severe). The area affected of each palm and sole is scored from 0 (0%) to 6 (90-100%). Scores for the 3 characteristics of PPP are summed and adjusted for the area affected, and the scores for each palm and sole are added to calculate the total score. The PPPASI total score ranges from 0 to 72. A higher score indicates more severe disease.
Time Frame: Baseline to Week 16
Population: Intent-to-treat analysis set with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Imsidolimab
Number analyzed (Participants) | 24 | 24
percentage of participants | 50.0 [29.12 to 70.88] | 45.8 [25.55 to 67.18]
Statistical Analysis 1: Comparison: Placebo vs Imsidolimab; Test type: Other; Odds Ratio (OR) = 0.879, 95% CI 2-sided [0.288 to 2.686] — Odds ratio from a logistic regression model including treatment as fixed effect, history of plaque psoriasis and Baseline PPPASI score as covariates and using multiple imputation for missing data

4. Secondary Outcome: Percentage of Participants Who Achieved a Clear or Almost Clear Palmoplantar Pustulosis Investigator's Global Assessment (PPPIGA) Score at Week 16
Description: The Investigator rated the severity of participants' disease on the following 5-point scale:
  * 0: Clear - No signs of palmoplantar pustulosis; no scaling or crusts or pustules remain;
  * 1: Almost clear - Slight scaling and/or erythema and/or slight crusts; very few (yellow) and/or old (brown) pustules;
  * 2: Mild - Scaling and/or erythema and/or crusts; visible new (yellow) and/or old (brown) pustules of limited number and extent;
  * 3: Moderate - Prominent scaling and/or erythema and/or crusting; prominent new (yellow) and/or old (brown) pustules covering most of the area involved;
  * 4: Severe - Severe scaling and/or erythema and/or crusting; numerous new (yellow) and/or old (brown) pustules with / without major confluence, covering the entire area of at least 2 palmoplantar sites.
Time Frame: Week 16
Population: Intent-to-treat analysis set with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Imsidolimab
Number analyzed (Participants) | 24 | 24
percentage of participants | 12.5 [2.66 to 32.36] | 20.8 [7.13 to 42.15]
Statistical Analysis 1: Comparison: Placebo vs Imsidolimab; Test type: Other; Odds Ratio (OR) = 2.6, 95% CI 2-sided [0.5 to 13.9] — Odds ratio from a logistic regression model including treatment as fixed effect, history of plaque psoriasis and Baseline PPPIGA score as covariates and using multiple imputation for missing data

ADVERSE EVENTS:
Time Frame: From first dose of any study drug to Week 24
Arm/Group | Placebo | Imsidolimab
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/30
Other Adverse Events (participants affected / at risk) | 20/29 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Imsidolimab (N=30)
Abortion early (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Imsidolimab (N=30)
Nasopharyngitis (Infections and infestations) | 4 | 4
Pharyngitis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Nerve compression (Nervous system disorders) | 0 | 1
Anosmia (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Panic attack (Psychiatric disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 5 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Blepharospasm (Eye disorders) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish trial results until after the first multi-center publication unless such publication is not published within a period that is at least 18 months but less than or equal to 24 months after trial completion. In addition, the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03633396/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03633396/SAP_001.pdf